CLINICAL TRIAL: NCT05063500
Title: A Multi-center, Randomized, Double-blind, Positive-controlled Phase Ⅲ Clinical Trial of Bicyclol Tablets in the Treatment of Acute Drug-induced Liver Injury
Brief Title: The Multi-Center, Randomized, Double-blind, Positive Controlled Clinical Trial of Bicyclol in the Treatment of Acute DILI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drug Induced Liver Disease Study Group (Other)
Collaborators: Beijing Union Pharmaceutical Factory Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHC-2020
Record Dates: First submitted 2021-09-09; First posted 2021-10-01 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Drug-Induced Acute Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — bicyclol; Tablets; polyene phosphatidylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group: each oral bicyclol 50mg, three times daily for 4 weeks.
  Interventions: Drug: bicyclol, 25mg/ tablet
- Control group (Active Comparator): Control group: each oral polyene phosphatidylcholine 456mg, three times daily for 4 weeks.
  Interventions: Drug: polyene phosphatidylcholine capsules, 228mg/ particle.

INTERVENTIONS:
Drug: bicyclol, 25mg/ tablet — Experimental group: each oral bicyclol 50mg, three times daily for 4 weeks.
  Arms: Experimental group
Drug: polyene phosphatidylcholine capsules, 228mg/ particle. — Control group: each oral polyene phosphatidylcholine 456mg, three times daily for 4 weeks.
  Arms: Control group

SUMMARY:
The study adopted the design of multi-center, randomized, double-blind, positive control drug, superiority test, using the double-blind double-simulating skills. The qualified subjects, according to the ratio of 1:1, were randomized into experimental group and positive drug control group and received a treatment course of 4 weeks, all individuals were followed up for 4 weeks after drug withdrawal.

DETAILED DESCRIPTION:
Further evaluated the safety and efficacy of bicyclol in the treatment of acute drug-induced liver injury using polyene phosphatidylcholine capsule as the positive control drug.

The study adopted the design of multi-center, randomized, double-blind, positive control drug, superiority test, using the double-blind double-simulating skills. The qualified subjects, according to the ratio of 1:1, were randomized into experimental group and positive drug control group and received a treatment course of 4 weeks, all individuals were followed up for 4 weeks after drug withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. 18~75 years old, male or female;
2. When screening, the threshold of serum liver biochemical test meets one of the following criteria: i: ALT≥5ULN; ii: ALP≥2ULN; iii: ALT≥3ULN, and TBiL≥2ULN;
3. During the screening, the patients with hepatocellular injury type or mixed type DILI mainly manifested by a significant increase in ALT were mainly selected;
4. Meeting the standard of clinical diagnosis of acute drug-induced liver injury, the RUCAM causality scale score is more than or equal to 6 points. If the RUCAM causality scale score is 3~5, the subject needs three liver disease experts to confirm whether he is DILI patient, meanwhile, at least two of three liver disease experts should have the same judgment.
5. Liver biochemical indexes (ALT, AST, ALP, GGT, TBiL, albumin, prothrombin time) abnormalities lasted no more than 90 days;
6. Patients can understand the nature of the experiment, the nature of the disease, the characteristic of drugs, related treatment methods, and the risk they may need to bear if they participate in the test and sign the informed consent.

Exclusion Criteria:

1. Liver injury is caused by other reasons, such as viral hepatitis, alcoholic liver disease, nonalcoholic fatty liver disease, etc.;
2. Patients with acute or subacute liver failure; patients with acute liver failure or liver decompensation, such as hepatic encephalopathy, ascites, albumin is less than normal value, International normalized ratio (INR) of prothrombin time greater than 1.5;
3. Cholestatic DILI;
4. Serum creatinine is more than 1.5 times ULN;
5. Severe or life-threatening heart, lung, brain, kidney, gastrointestinal and systemic diseases;
6. Simultaneous application of drugs that affect the efficacy of this trial;
7. Allergy or intolerance to experimental drugs;
8. With no ability to express their complaints, such as mental illness and severe neurosis patient;
9. The patient can not cooperate and poor compliance;
10. Pregnant and lactating women or women preparing for pregnancy;
11. The patient participated in other clinical trials in 3 months before entering this study;
12. Using other liver-protective drugs except ursodeoxycholic acid or ademetionine within last 3 days;
13. The researchers consider not suitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The normalization rate of serum ALT after 4 weeks of treatment | After 4 weeks of treatment
  The normalization rate of serum ALT after 4 weeks of treatment

SECONDARY OUTCOMES:
The normalization rate of serum ALT after 2 weeks of treatment | After 2 weeks of treatment
  The normalization rate of serum ALT after 2 weeks of treatment
The decrease value in serum ALT relative to baseline at 2 weeks of treatment; | After 2 weeks of treatment
  The decrease value in serum ALT relative to baseline at 2 weeks of treatment;
The decrease value in serum ALT relative to baseline at 4 weeks of treatment; | After 4 weeks of treatment
  The decrease value in serum ALT relative to baseline at 4 weeks of treatment;
The time from the start of treatment to the return of ALT | Up to 4 weeks
  The time from the start of treatment to the return of ALT
The normalization rate of serum AST after 2 weeks of treatment | After 2 weeks of treatment
  The normalization rate of serum AST after 2 weeks of treatment
The normalization rate of serum AST after 4 weeks of treatment | After 4 weeks of treatment
  The normalization rate of serum AST after 4 weeks of treatment
The decrease in serum AST relative to baseline at 2 weeks of treatment. | After 2 weeks of treatment
  The decrease in serum AST relative to baseline at 2 weeks of treatment.
The decrease in serum AST relative to baseline at 4 weeks of treatment. | After 4 weeks of treatment
  The decrease in serum AST relative to baseline at 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Mao, Study Chair — RenJi Hospital; Chengwei Chen, Study Chair — 905th Hospital of Pla Navy
Locations (2):
- China (2):
  - Renji Hospital ，Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - 905th Hospital of Pla Navy, Shanghai, Shanghai Municipality